CLINICAL TRIAL: NCT06419842
Title: Evaluation of the Impact of Hypnosis for Performing Lumbar Infusion Tests.
Brief Title: Impact of Hypnosis for Performing Lumbar Infusion Tests
Acronym: HYPNINF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: PI2023_843_0149
Record Dates: First submitted 2024-05-14; First posted 2024-05-17 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Hypnosis; Hydrocephalus; Anxiety; Pain
Keywords: hypnosis; infusion study; Hydrocephalus; Anxiety; Pain
MeSH Terms: conditions — Hydrocephalus; Anxiety Disorders; Pain | interventions — Hypnosis; methyl hydroxyethyl cellulose

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- hypnosis (Experimental): In group 1, the patient benefits from a dedicated nurse consultation. During this consultation, the nurse will explain the highlights of the hospitalization, the procedure and anticipate the hypnosis technique to be used. The technique chosen during the consultation will be applied during the test. The nurse is positioned at the head of the patient and with physical contact.
  Interventions: Other: hypnosis
- comfort (Sham Comparator): In group 2, the patient benefits from a nurse consultation. Non-medicinal techniques are not offered. During the infusion test, the nurse will be positioned at the patient's head allowing proximity but without oral or physical intervention.
  Interventions: Other: comfort
- standard (No Intervention): In group 3, the IDE consultation is performed according to the same modalities as in group 2. During the procedure, the nurse will be out of the patient's field of vision and will assist the surgeon in the installation behind the patient. Only the surgeon will interact with the patient.

INTERVENTIONS:
Other: hypnosis — the patient benefits from a dedicated nurse consultation. During this consultation, the nurse will explain the highlights of the hospitalization, the procedure and anticipate the hypnosis technique to be used. The technique chosen during the consultation will be applied during the test. The nurse is positioned at the head of the patient and with physical contact.
  Arms: hypnosis
Other: comfort — the patient benefits from a nurse consultation. Non-medicinal techniques are not offered. During the infusion test, the nurse will be positioned at the patient's head allowing proximity but without oral or physical intervention.
  Arms: comfort

SUMMARY:
Infusion tests are now the gold standard for the diagnosis of chronic adult hydrocephalus (CAH), also known as normal pressure hydrocephalus. It is an invasive procedure using the same approach as a lumbar puncture. Once the intrathecal puncture is performed, the intracranial pressure is measured in lateral decubitus via a pressure head. Dynamic tests (injection of 0.9% NaCl at a constant flow rate) are performed after recording the basal pressure. This type of test lasts 30 to 45 minutes in lateral decubitus. Patients with CAH have cognitive-behavioral disorders that can alter the gesture and its interpretation in case of movements or contractures. Movement artefacts lead to a longer recording time. The longer the test, the more the patients' tolerance tends to decrease. Moreover, the patient's feeling towards this test is important because it may have to be repeated. Pain, anxiety and patient comfort are essential parameters to consider. Non-medicinal techniques (hypnosis, music therapy) have shown a tendency to reduce anxiety in pediatric and adult populations with an impact on instantaneous anxiety but also on personality-related anxiety. Most studies are focused on specific pathologies, primarily in palliative care, or on pediatric application. The use of these techniques in an elderly population with mild cognitive-behavioral disorders has not been explored.

The objective is to evaluate the impact of hypnosis on anxiety, pain and comfort during the lumbar infusion test.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 65 years old undergoing assessment for suspected CAH in day hospitalization for a lumbar infusion test
* No major cognitive impairment (MMSE>20)

Exclusion Criteria:

* Patient less than 65 years old
* Major cognitive impairment (MMSE<20)
* History of lumbar surgery
* Contraindication to lumbar puncture or infusion test
* Hearing impairment

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-05-14 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Decrease in anxiety in group 1compared to the other groups | 2 years
  Decrease in anxiety in group 1 compared to the other groups

SECONDARY OUTCOMES:
Decrease in pain in group 1 | 2 years
  Decrease in pain on the numerical scale in group 1 versus other groups
Increase in comfort in group 1 | 2 years
  Increase in comfort on the numerical scale in group 1 versus the other groups
Better overall patient impression in group 1 versus other groups | 2 years
  Better overall patient impression (Likert scale) in group 1 versus other groups
Less heart rate variation in group 1 versus other groups | 2 years
  Less heart rate variation in group 1 versus other groups
Decreased puncture time required in group 1 versus other groups | 2 years
  Decreased puncture time required in group 1 versus other groups
fewer position changes required in group 1 versus other groups | 2 years
  fewer position changes required in group 1 versus other groups

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens Picardie, Amiens, Picardie, France

IPD SHARING:
Plan to Share IPD: No